CLINICAL TRIAL: NCT03975946
Title: Efficacy and Tolerance of RHEOpheresis in the Treatment of Peripheral Artery Disease in Hemodialysis Patients: a Prospective Randomized Single-blind Trial
Brief Title: Efficacy and Tolerance of RHEOpheresis in the Treatment of Peripheral Artery Disease in Hemodialysis Patients
Acronym: RHEO-PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-68; 2019-A01513-54 (Other: ID RCB); RCAPHM18_0384 (Other: AP-HM)
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The efficacy will be assessed by a vascular surgeon blinded to the study group during consultation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the rheopheresis group (Active Comparator)
  Interventions: Procedure: Rheopheresis procedure; Biological: Blood Sample
- the shamapheresis group (Placebo Comparator)
  Interventions: Biological: Blood Sample; Procedure: Shamapheresis procedure

INTERVENTIONS:
Procedure: Rheopheresis procedure — Rheopheresis is performed using an automated monitor in a double-filtration cascade. Plasma purify from of high molecular weight proteins through a secondary filter is then returned to the patient. This technique is performed in tandem with a hemodialysis monitor.
  Arms: the rheopheresis group
Biological: Blood Sample — Biological analysis
Procedure: Shamapheresis procedure — Shamapheresis is performed with the same automated monitor (Plasauto, HemaT company). Extracted plasma is not treated through the secondary filter (Rheofilter) and return to the patient. This technique is performed in tandem with a hemodialysis monitor.
  Arms: the shamapheresis group

SUMMARY:
Peripheral arterial disease (PAD) with limb-threatening ischemia (PAD-LTI) involves both macrocirculation and microcirculation. Macrocirculatory abnormalities are accessible to revascularization techniques (endovascular or surgical) contrary to microcirculatory abnormalities. Conservative treatments have limited efficacy in patients with end-stage renal disease (ESRD). There is no alternative treatment for patients with PAD-LTI in hemodialysis.

Rheopheresis is an apheresis technique specifically designed for the treatment of microcirculatory disorders in which anomalies of rheology are at the center of physiopathology. This double cascade plasma filtration technique reduces plasma viscosity and eliminates inflammation mediators which play an essential role in PAD. This technique has already shown its effectiveness in a randomized trial in dry Age-related macular degeneration (AMD), another pathology of microcirculation. The effectiveness of rheopheresis in PAD-LTI has only been reported in a small number of cases.

This Hypothesis is that the treatment of microcirculation by rheopheresis would improve wound healing of the ischemic lesion and/or reduce major amputation and thus the prognosis of the affected limb of the patient with PAD-LTI in hemodialysis. This objective is to demonstrate the efficacy of rheopheresis, (twelve sessions), to avoid major amputation and reaches complete wound healing of ischemic lesion in the dialysis patient population with PAD-LTI. This study is prospective, Controlled, Parallel, Randomized, Single blind and Multicentric in France (12 French centers).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* End stage renal disease (ESRD) treated by hemodialysis or hemodiafiltration
* PAD-LTI with tissue loss and/or wounds (ulcers or gangrene) with at least one of the following criterion: arterial pressure assessment at the ankle <70 millimeter of mercury (mmHg), or toe pressure 30 mmHg, or transcutaneous oximetry measurements < 40 mmHg
* Interventional or surgical revascularization either not technically possible or no necessary. Or if revascularization has already been performed and the diagnosis of chronic critical ischemia is maintained.
* Female of childbearing potential, will have to use highly effective methods of contraception from study start to the end.
* Medical insurance
* Signed informed consent

Exclusion Criteria:

* Need for revascularization either endovascular (angioplasty) or surgery (bypass) of the ischemic lesion area
* Pregnancy or breastfeeding and all the other categories of people with special protection according to the French Code de la Santé Publique (CSP): patients under legal supervision, patients hospitalized without contentment, patients admitted in social or sanitary structures for care and not research, and patients in emergency situations
* Uncontrolled infection (persistence of fever despite appropriate antibiotic therapy)
* Life expectancy greater than 1 year
* Severe cognitive or psychiatric disorders
* History of allergic reaction to dialysis membrane
* Patients unable to give an informed consent or unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of complete wound healing of the ischemic lesions | 8 months
  Complete wound healing will be assessed clinically by complete epithelialization of the ischemic lesion
Percentage of absence of major amputation. | 8 months
  Major amputation will be defined as above-the-knee amputation (AKAs) and below-the-knee amputation above the ankle (BKAs)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No